CLINICAL TRIAL: NCT01369368
Title: Treatment of Relapsed Acute Leukemia After Allogeneic Stem Cell Transplantation: Disease Stabilization Through Chemotherapy, Immunomodulatory Treatment and Immunotherapy
Brief Title: Treatment of Acute Leukemia Relapse After Allotransplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Øystein Bruserud, Professor, University of Bergen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allo-Relapse-2011
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Allogeneic stem cell transplantation; Relapse; Disease stabilization, survival
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Azacitidine, valproic acid, all-trans retinoic acid, hydroxyurea, eventually donor leukocyte infusions
  Interventions: Drug: Combined use of azacitidine, valproic acid, hydroxurea and eventually donor leukocyte infusions.

INTERVENTIONS:
Drug: Combined use of azacitidine, valproic acid, hydroxurea and eventually donor leukocyte infusions. — Azacitidine 100 mg day 1-3 in each cycle Valproic acid, continuous therapy from day 1 All-trans retinoic acid 22.5 mg/m2 twice daily day 1-14 in each cycle Hydroxurea 500 mg initially eventually increased to 1 g daily. Eventually donor leukocyte infusions on day 10 from the second cycle.
  Other Names: Give as repeated cycles with 5 weeks intervals. Donor leukocyte infusions are allowed from cycle 2.

SUMMARY:
Patients with relapse of acute leukemia often only receive supportive therapy. Our hypothesis is that a combination therapy can stabilize the disease for patients with early relapse after allogeneic stem cell transplantation. The investigators will combine 5-azacitidine 100 mg daily subcutaneously (days 1-3), valproic acid (continuous therapy from day 1), All-trans retinoic acid (days 1-14) and hydroxurea (continuous treatment from day 15 of first cycle. Azacitidine and ATRA can be repeated with 5 weeks intervals, donor leukocyte infusions on day 10 is allowed from the second cycle.

ELIGIBILITY:
Inclusion Criteria:

* AML relapse within one year after transplantation
* Blood and marrow sampling being possible
* Expected survival at least 4 weeks
* No expected drug interactions
* Informed consent possible

Exclusion Criteria:

* Intolerance to any study drug
* Serious kidney or liver disease
* Informed consent not possible
* Previous pancreatitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Disease stabilization | 5 years
  Strict criteria defined in the protocol.

SECONDARY OUTCOMES:
Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway